CLINICAL TRIAL: NCT05819905
Title: Prediction of Lung Cancer Characteristics Using PET/CT Radiomics
Brief Title: Radiomics for prEdiction of lunG cAncer biologY
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REGAL
Record Dates: First submitted 2023-03-17; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Non Small Cell Lung Cancer; PET/CT; PD-L1; Gene Mutation-Related Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT — Pre treatment staging 18F-FDG PET/CT

SUMMARY:
Therapeutic progress for subgroups of Non Small Cell Lung Cancer can largely be attributed to the accumulation of molecular knowledge and the development of new drugs that specifically target molecular abnormalities. An understanding of the immune landscape of tumors, including immune-evasion strategies, has also led to breakthrough therapeutic advances.These new options require prior treatment tumoral sampling to identify patients who have neoplasms with specific genomic aberrations or favorable immune environment. Medical imaging and radiomic approach may provides surrogate markers non invasively.The objective of the present retrospective study is to build and validate a predictive model of common molecular alterations and PD-L1 expression in NSCLC using pre treatment PET/CT derived radiomics.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NSCLCC
* pre treatment 18F FDG PET/CT
* available molecular biology and histology results

Exclusion Criteria:

* non available PET/CT images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically proven NSCLC with molecular biology analysis and initial staging PET/CT
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
prediction of PDL1 expression | 1 month
  Evaluation of the performances of PET/CT derived radiomics to predict PDL1 expression >1% (PDL1 : Programmed death-ligand 1 as previously determined on routine tumoral biopsy): area under the receiver operating characteristics curve (AUC), accuracy, sensitivity and specificity.
prediction of EGFR genomic alteration | 1 month
  Evaluation of the performances of PET/CT derived radiomics to predict the presence of EGFR mutation (EGFR: epidermal growth factor receptor, presence /or not of EGFR alteration as previously determined on routine tumoral biopsy): area under the receiver operating characteristics curve (AUC), accuracy, sensitivity and specificity.

SECONDARY OUTCOMES:
Prediction of KRAS alteration | 1 month
  Evaluation of the performances of PET/CT derived radiomics to predict the presence of KRAS mutation (KRAS : Kirsten rat sarcoma viral oncogene : presence/or not of KRAS alteration as previously determined on routine tumoral biopsy): area under the receiver operating characteristics curve (AUC), accuracy, sensitivity and specificity.
Prediction of BRAF mutation | 1 month
  Evaluation of the performances of PET/CT derived radiomics to predict the presence of BRAF mutation (BRAF : raf murine sarcoma viral oncogene homolog B, presence/or not of BRAF mutation as previously determined on routine tumoral biopsy): area under the receiver operating characteristics curve (AUC), accuracy, sensitivity and specificity.
Prediction of ALK/ROS translocation | 1 month
  Evaluation of the performances of PET/CT derived radiomics to predict the presence of ALK/ROS translocation (ALK : anaplastic lymphoma receptor tyrosine kinase, ROS : c-ROS protooncogene 1; presence /or not of ALK and ROS alteration as previously determined on routine tumoral biopsy): area under the receiver operating characteristics curve (AUC), accuracy, sensitivity and specificity.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Poitiers, Poitiers, France